CLINICAL TRIAL: NCT01008592
Title: The Effect of Levocetirizine (Xyzal®) on the Skin Levels of Inflammatory Mediators Histamine, Serine Proteases, Prostaglandin E2, Leukotriene B4 and Cathepsins in Patients With Symptomatic Dermatographism and Chronic Idiopathic Urticaria
Brief Title: The Effect of Levocetirizine on Inflammatory Mediators in Dermatographism
Status: Terminated | Type: Observational
Why Stopped: Mediators of interest were not consistently detectable with the analytical methods employed.
Sponsor: Wake Forest University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: GTS# 33519
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2009-11

CONDITIONS: Rhinitis; Urticaria
Keywords: dermatographism, levocetirizine (Xyzal); chronic idiopathic urticaria, dermatographism
MeSH Terms: conditions — Rhinitis; Urticaria; Familial dermographism; Chronic Urticaria | interventions — levocetirizine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Subjects with chronic idiopathic urticaria exhibiting dermatographism.
  Interventions: Drug: levocetirizine or placebo

INTERVENTIONS:
Drug: levocetirizine or placebo — oral administration, single tablet, 5 mg.
  Other Names: Xyzal

SUMMARY:
Levocetirizine (Xyzal®), the active levorotatory enantiomer of cetirizine (Zyrtec®), is a FDA-approved drug used in the treatment of symptoms associated with seasonal and perennial allergic rhinitis and chronic idiopathic urticaria. The parent compound, cetirizine was shown to be effective against experimental dermatographism, however no study has been conducted so far on the effect of levocetirizine on the inhibition of dermatographism. It is known that cetirizine is a mast-cell stabilizer and decreases histamine levels and the number of tryptase positive mast cells. Cetirizine inhibits the production of interleukin 8 (IL8) and leukotriene B4 (LTB4) by immune cells - two potent chemoattractants - and induces the release from monocytes of prostaglandin E2 (PGE2), a suppressor of antigen presentation and MHC class II expression. However, the effects of the most active enantiomer levocetirizine on these inflammatory mediators have not been evaluated so far. Therefore, we aim to conduct a study in humans with dermatographism and chronic idiopathic urticaria to evaluate the effect of levocetirizine on the above-mentioned mediators. The study will involve the use of skin microdialysis, a minimally invasive technique to measure inflammatory mediators in the extracellular space in dermis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic dermatographism and chronic idiopathic urticaria.
2. Adult male and female between 18 to 60 years of age.
3. Signature of informed consent.
4. No known hypersensitivity to levocetirizine or to any of the ingredients of Xyzal® or to cetirizine.
5. Willingness to refrain from other antihistamines, prescription and and over- the-counter cough & cold medications, topical creams, topical steroids and topical immunomodulators, for one week prior to the study. In very severe cases of CIU and dermatographism, based on dermatologist consultation and recommendation, and depending on the half-life of the prior antihistamine medication used, this period may be reduced to 3-4 three days. Rescue medication will be promptly provided if at any time the subjects will experience a significant relapse of their CIU symptoms.
6. Good general health.
7. Ability to understand and comply with the protocol.
8. Females of child-bearing potential must have a negative urine pregnancy test prior to randomization.
9. Absence of another active skin disease that may influence skin evaluation during the study.

Exclusion Criteria:

1. Pregnant females, females planning on getting pregnant or breast feeding.
2. Uncontrolled chronic disease such as diabetes.
3. The presence of renal disease with a moderate or severe renal impairment (since Xyzal is primarily eliminated through the kidneys) as documented from medical records or patient history.
4. History of anaphylaxis, angioedema or allergy to Xyzal or cetirizine (Zyrtec).
5. Any systemic disease involving mast cells such as allergic rhinitis, lung disease, asthma or autoimmune collagen disease.
6. Severe vascular or neurological diseases that would impart an asymmetric blood perfusion or an impaired function of the arms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study subjects will be adult patients with dermatographism and chronic idiopathic urticaria from the Wake Forest University Health Sciences Dermatology Clinic population and patients recruited via appropriate IRB-approved advertising. Subjects will show definitive clinical findings compatible with dermatographism and chronic idiopathic urticaria as assessed by one of the investigators. Twenty subjects with dermatographism and chronic idiopathic urticaria will be recruited. Eligible subjects will include adult men and women 18 to 60 years of age with chronic disease.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the inhibitory effect of levocetirizine in the induction of dermatographism. To assess the levels of key inflammatory mediators and proteases in the skin during dermatographic reaction, using microdialysis. | Time-points are selected within a 5 hours interval, during experimental microdialysis

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Department of Dermatology, Winston-Salem, North Carolina, United States